CLINICAL TRIAL: NCT01445223
Title: A Study on ART Naïve Patients On Different Regimens to Treat Hiv (a Phase 4 Study)
Brief Title: A Study on Antiretroviral Therapy (ART) Naïve Patients On Different Regimens to Treat Hiv (NORTHIV)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Göteborg University (Other)
Responsible Party: Principal Investigator, Lars-Magnus Andersson, Principal Investigator, Göteborg University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Northiv protocol 3.66
Record Dates: First submitted 2011-09-28; First posted 2011-10-03 (Estimated); Last update posted 2011-10-04 (Estimated); Status verified 2011-10

CONDITIONS: HIV
Keywords: HIV; Antiretroviral therapy; efavirenz; lopinavir; atazanavir; randomised controlled clinical trial
MeSH Terms: interventions — Lopinavir; atazanavir, ritonavir drug combination; efavirenz

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- lopinavir/ritonavir (Active Comparator): 400/100 mg BID + 2 NRTIs BID
  Interventions: Drug: Lopinavir ritonavir
- atazanavir/ritonavir (Active Comparator): 300mg+100mg QD+ 2 NRTI QD
  Interventions: Drug: Atazanavir ritonavir
- efavirenz (Active Comparator): 600mg QD + 2NRTI QD
  Interventions: Drug: Efavirenz

INTERVENTIONS:
Drug: Lopinavir ritonavir — 400mg BD 100mg BD
  Arms: lopinavir/ritonavir
Drug: Atazanavir ritonavir — 300mg QD 100mg QD
  Arms: atazanavir/ritonavir
Drug: Efavirenz — 600mg QD
  Arms: efavirenz

SUMMARY:
The present study aims to compare efficacy, side-effects, and treatment adherence of three different treatment regimens given to antiretroviral naïve HIV-1 infected patients. Treatment will be initiated in accordance with the Swedish National Guidelines. In the twice daily (BID) arm (1), which could be considered as a standard regimen at present, lopinavir/ritonavir, is co-administrated with 2 nucleoside reverse transcriptase inhibitors (NRTIs) administrated BID. The first once daily (QD) arm (2) combines the protease inhibitor (PI) atazanavir/ritonavir with 2 NRTIs administrated QD, and in the second QD arm (3), the non nucleoside reverse transcriptase inhibitor (NNRTI) efavirenz is combined with 2 NRTIs administrated QD. All drugs used in the study are licensed in the participating countries and patients will be followed as in clinical practice. Patients could optionally, after informed consent, be followed with additional measurements of HIV-1 RNA after 1, 2, and 3 weeks of treatment to asses the kinetics of viral decline after initiation of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 16 years of age
* HIV-1 infected as documented by a licensed HIV-1 antibody ELISA
* Ability to understand and provide informed consent
* Indication for antiretroviral treatment
* Antiretroviral naïve
* All clinical laboratory values not clinically significant

Exclusion Criteria:

* Subjects being pregnant
* Women of childbearing potential not practicing birth control
* Subjects with renal failure requiring dialysis
* Drug interactions with any of the study drugs that are not manageable
* Resistance to any of the study drugs

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2004-04; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Intention to treat (ITT)/time to loss of virological response (TLOVR) | 144 weeks
  1. Virological failure (see 5.5.2 for definition)
  2. Treatment interruption or change of study treatment due to side-effects
  3. Treatment interruption or change of study treatment due to any other reason
  4. Missed to follow-up
  1. HIV-1 RNA >50 copies/ml in two consecutive measurements from week 24 and on 2. any rise in HIV-1 RNA >50 copies/ml in two consecutive measurements after viral load <50 copies/ml has been reached 3. HIV-1 RNA never <50 copies/ml after week 24

SECONDARY OUTCOMES:
Frequency of abnormal laboratory parameters | 144 weeks
  Incidence of abnormal laboratory parameters at follow-up
Adherence to study medication | 144 weeks
  Proportion of doses taken correctly
Frequency of adverse events | 144 weeks
  Proportion of treatment discontinuations and changes due to different adverse events
Changes in CD4 cell counts | 144 weeks
  Changes in CD4+ T-cell count from baseline
Changes in plasma lipids | 144 weeks
  Changes from baseline in plasma lipids
Frequency of hyperlipidemia | 144 weeks
  Incidence of hypercholesterolemia and hypertriglyceridemia at baseline and follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Magnus Gisslén, Professor, Principal Investigator — Goteborg Universitet
Locations (1):
- Department of Infectious Diseases, Gothenburg, Goteborg, Sweden

REFERENCES:
- [Result] Eden A, Andersson LM, Andersson O, Flamholc L, Josephson F, Nilsson S, Ormaasen V, Svedhem V, Sall C, Sonnerborg A, Tunback P, Gisslen M. Differential effects of efavirenz, lopinavir/r, and atazanavir/r on the initial viral decay rate in treatment naive HIV-1-infected patients. AIDS Res Hum Retroviruses. 2010 May;26(5):533-40. doi: 10.1089/aid.2009.0177. PMID 20455766
- [Result] Josephson F, Andersson MC, Flamholc L, Gisslen M, Hagberg L, Ormaasen V, Sonnerborg A, Vesterbacka J, Bottiger Y. The relation between treatment outcome and efavirenz, atazanavir or lopinavir exposure in the NORTHIV trial of treatment-naive HIV-1 infected patients. Eur J Clin Pharmacol. 2010 Apr;66(4):349-57. doi: 10.1007/s00228-009-0763-z. Epub 2009 Dec 5. PMID 19967342
- [Derived] Vesterbacka J, Nowak P, Barqasho B, Abdurahman S, Nystrom J, Nilsson S, Funaoka H, Kanda T, Andersson LM, Gisslen M, Sonnerborg A. Kinetics of microbial translocation markers in patients on efavirenz or lopinavir/r based antiretroviral therapy. PLoS One. 2013;8(1):e55038. doi: 10.1371/journal.pone.0055038. Epub 2013 Jan 28. PMID 23383047
- See also: Goteborg University — http://www.sahlgrenska.gu.se/